CLINICAL TRIAL: NCT05886738
Title: Investigating the Effect of Short-term Fasting on T Cell Metabolism, Function, and Phenotype in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Dr. Jonathan Little, Principle Investigator, Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H22-03605
Record Dates: First submitted 2023-05-12; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Fasting; T-Cell Dysfunction
MeSH Terms: conditions — Obesity; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Masking Description: Participants will be fasting for 48 hours so it will not be possible to mask the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese (Experimental): Individuals with obesity will be recruited. Obesity will be defined as having a body mass index >= 30 kg/m2 or a waist circumference of > 88cm (females) or >102 cm (males).
  Interventions: Other: Fasting
- Lean (Active Comparator): Lean individuals will be recruited and will act as the reference arm such that we will compare responses of individuals with obesity to the lean group. This group will be defined as having a BMI between 18.5-24.9 kg/m2 and a waist circumference of less than 88 cm (females) or 102 cm (males)
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — Obese and lean groups will fast for 48 hours, followed by a 3-hour refeeding period.

SUMMARY:
The immune system is made up of many types of immune cells, each of which play a specialized role in protecting against pathogens. T cells are a crucial part of the adaptive immune system, and receive signals from the body's metabolism which tell them whether they should become activated to respond to an infection or if they should stay in their resting state. In obesity, the body's metabolism shifts and these T cells become less effective at protecting against infection and instead start to increase inflammation which is involved in obesity-related health conditions. The investigators are conducting this study because the investigators are interested in understanding how fasting, which will alter the metabolic signals that T cells receive, might impact the types of T cells that are present and how they respond to activating signals. Additionally, the investigators are interested in understanding if these responses differ between T cells from individuals with obesity versus lean individuals.

DETAILED DESCRIPTION:
Recruitment and Eligibility:

This is a two-group pre-post study which has been approved by the UBC Clinical Research Ethics Board (H22-03605). Participants will be recruited from the community and the UBC Okanagan campus with posters and social media posts. Additionally, an email invitation will be sent to participants from past studies that have indicated on their previous Consent Forms that they agree to be contacted for future research studies. The investigators will aim to recruit equal numbers of males and females in each group. Interested volunteers will be initially screened via a standardized phone call to determine if they meet the eligibility criteria. If the eligibility criteria are met, they will be invited to participate in the study, researchers will discuss the study details with the potential participant, and participants will be sent the Consent Form to review and sign if they consent to participate. This study will compare the responses of individuals with obesity to individuals that are lean. Lean individuals will be included if they have a body mass index (BMI) between 18.5 and 24.9 kg/m2 and a waist circumference < 88 cm (females) or < 102 cm (males). Individuals with obesity will be included if they have a BMI of > 30 kg/m2 or a waist circumference > 88 cm (females) or > 102 cm (males). Lean individuals will be age- and sex-matched to individuals with obesity, and individuals in both groups will be included if they are 19-69 years of age and are physically inactive. This will be defined as accumulating < 150 minutes of moderate-to-vigorous physical activity per week or participating in moderate-to-vigorous physical activity < 3 days per week. Additionally, all participants must be able to read and understand English in order to complete the study diet logs. Interested volunteers will be excluded if they have a diagnosed autoimmune or inflammatory disease, have had a cancer diagnosis and/or treatment within the last 5 years, diagnosed type 1 or 2 diabetes, or a history of cardiovascular events (i.e., heart attack, stroke), and/or are currently pregnant. Additionally, interested volunteers will be excluded if they take glucose-lowering or thyroid medications, or if they currently smoke cigarettes or cannot refrain from smoking/using cannabis for the duration of the study. Finally, individuals that actively take ketone supplements, practice intermittent fasting with regular periods of fasting > 24 hours, follow a ketogenic diet, or are actively trying to lose or gain weight (> 4 kg weight loss or gain in last month) will be excluded from the study.

Visits Summary This study will involve a total of 3 visits across 48 hours during which participants will be in the laboratory for a total of 5 hours (study design pictured in Figure 1). Participants will be fasted during the 48 hours, and upon arrival to their final visit will be provided with a meal.

Prior to coming in to the lab the investigators will have already obtained informed consent, and the investigators will have participants log all of the food and drinks that they consume in a diary for the 3 days before their first visit. They will bring this 3-day food log with them to their first visit to the lab. Additionally, the investigators will ask participants not to consume any alcohol or participate in any exercise the day before their first visit.

Visit 1: 1 hour On the first visit, participants will consume a standardized breakfast (meal replacement drink). Once they have consumed this meal, their fast will begin and they will arrive at the laboratory 4 hours later. Researchers will measure height, body weight, waist circumference, and blood pressure. A blood sample will be obtained from the antecubital vein by a trained phlebotomist (Hashim Islam, PhD; Helena Neudorf, PhD student) using a standard 21-gauge needle. Approximately 20 ml of blood will be drawn into EDTA tubes. Following this, the investigators will measure resting metabolic rate (RMR). To do this, participants will rest lying down in a supine position and connected to a metabolic cart (Parvo Medics TrueOne 2400) with which their expired air will be collected and analyzed for 30 minutes. Participants will be instructed not to consume any food or beverages other than water or calorie- and sugar-free beverages (provided by the researchers) if they wish, or partake in any moderate-to-vigorous physical activity for the duration of their fast.

Visit 2: 30 minutes Participants will arrive for their second visit 24 hours following their first visit. During this visit, 20 ml of blood will be obtained by a trained phlebotomist in the same manner as the first visit, and participants will again be offered calorie- and sugar-free beverages if they wish.

Visit 3: 3.5 hours Participants will arrive for their third and final visit having fasted for 48 hours. RMR and a blood sample (20 ml) will be collected, and participants will be provided with the same meal replacement drink a standardized breakfast to end their fast. Participants will remain in the laboratory for the next 3 hours, during which the investigators will collect RMR on the second half of every hour in the same manner as the first visit. At the end of the 3 hours, the investigators will collect a final blood sample (20 ml) will be collected.

Statistical Analyses Changes in all variables over time will be compared between the two groups using a linear mixed effects model with subject included as a random factor and group, time, and baseline measures will be included as fixed factors.

ELIGIBILITY:
Inclusion Criteria:

1. are 19-69 years of age, and
2. have body mass index (BMI) of between 18.5 and 24.9 kg/m2 and a waist circumference of less than 88 cm (females) or 102 cm (males), or
3. have a BMI over 30 kg/m2 or a waist circumference of more than 88 cm (females) or 102 cm (males)
4. can read and understand English

Exclusion Criteria:

1. Have a diagnosed autoimmune or inflammatory disease
2. Have had a cancer diagnosis and/or treatment within the last 5 years
3. Have diagnosed type 1 or 2 diabetes
4. Have a history of cardiovascular events (e.g., heart attack, stroke)
5. Are taking glucose-lowering or thyroid medications
6. Are currently taking ketone supplements, practice intermittent fasting, following a ketogenic diet, or are actively trying to lose or gain weight (more than 4 kg weight loss or gain in the last month)
7. Are accumulating 150 minutes or more of moderate-to-vigorous physical activity per week, or are participating in moderate-to-vigorous physical activity on 3 or more days per week
8. Smoke cigarettes or cannot refrain from smoking/using cannabis for the duration of the study
9. Are currently pregnant

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the rate of T cell fat-supported oxidative mitochondrial respiration assessed by Oroboros O2K after 48 hours of fasting | Baseline and 48 hours
  T cell respiration will be characterized in inactivated and activated T cells collected at baseline and after 48 hours of fasting. Inactivated T cells will be assessed immediately following isolation. Activated T cells will be assessed after culturing with CD3/CD28 for 24 hours.

SECONDARY OUTCOMES:
Change from baseline in the frequency (%) of T cell subsets assessed by multi-colour flow cytometry | Baseline and 48 hours
  Isolated T cells collected at baseline and after 48 hours of fasting will be cultured with CD3/CD28 for 24 hours after which their phenotype will be assessed to determine the frequency (%) of the major T cell subsets. The T cell subsets that will be characterized are T regulatory cells, subsets of T helper cells (Th1, Th2, Th17, Th22), and subsets of cytotoxic T cells (Tc1, Tc2, Tc17, and Tc22).
Change from baseline in the rate of T cell proliferation assessed by cell number | Baseline and 48 hours
  Isolated T cells collected at baseline and after 48 hours of fasting will be cultured with CD3/CD28 for 72 hours. The rate of cell proliferation after 72 hours is indicative of T regulatory cell suppressor function.

REFERENCES:
- [Derived] Sandilands RE, Neudorf H, Ursel S, Shaba H, Barg D, Vaz E, Schimweg P, Islam H, Little JP. Metabolic responses to 48-hour fasting and refeeding in adults with and without obesity. Appl Physiol Nutr Metab. 2026 Feb 6. doi: 10.1139/apnm-2025-0447. Online ahead of print. PMID 41650389
- [Derived] Neudorf H, Sandilands RE, Ursel S, Shaba H, Barg D, Tsusaka T, Moya-Garzon MD, Vaz E, Schimweg P, Goldberg EL, Long JZ, Kruger K, Islam H, Little JP. Altered immunometabolic response to fasting in humans living with obesity. iScience. 2025 Jun 11;28(7):112872. doi: 10.1016/j.isci.2025.112872. eCollection 2025 Jul 18. PMID 40662191